CLINICAL TRIAL: NCT06384001
Title: Mindfulness-based Meditation for Older Adults With Chronic Low Back Pain Based on the Gut-brain Axis: A Pilot Randomized Controlled Trial
Brief Title: Meditation for Older Adults With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jie Chen, PhD, RN, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004032
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low Back Pain
Keywords: Mindfulness; Older adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active MBM (Experimental): The active MBM is designed to be applied for 20 minutes per session daily.
  Interventions: Behavioral: Active MBM
- Sham MBM (Sham Comparator): The sham MBM intervention matches the active MBM
  Interventions: Behavioral: Sham MBM

INTERVENTIONS:
Behavioral: Active MBM — The MBM is designed to be applied for 20 minutes per session daily for two weeks. The recording will instruct participants to close their eyes, connect to the openness of one's minds, and mindfully maintain and deepen the connection through breathing with more openness and awareness. The MBM intervention will include three recordings that gradually take the participant into a more profound meditation practice. Participants will be instructed to listen to Meditation 1 for the first three days of the intervention, then switch to Meditation 2 for days 4-6 and Meditation 3 for the remainder of the 2-week intervention. The participants will be asked to practice meditation for eight weeks (6 weeks after the initial two weeks of MBM practice).
  Arms: Active MBM
Behavioral: Sham MBM — The sham MBM intervention was also recorded. The sham recording will instruct participants to relax and take deep breaths every 3 minutes without the specific mindfulness-based instructions (e.g., practicing mindful attention to the breath in a non-evaluative manner). All other aspects of the sham MBM intervention (e.g., body position, time spent listening to instructions, eyes closed) will match the active MBM.
  Arms: Sham MBM

SUMMARY:
This pilot randomized controlled trial aims to recruit 66 community-dwelling older adults with chronic low back pain and follow up them for 8 weeks. This study aims to test the preliminary effect of a mindfulness-based meditation (MBM) intervention on pain and symptoms among community-dwelling older adults with chronic low back pain, and also to test the effect of the MBM intervention on the host Gut-Brain Axis (GBA).

DETAILED DESCRIPTION:
Aim 1: to test the preliminary effect of a mindfulness-based meditation (MBM) intervention on pain and symptoms among community-dwelling older adults with chronic low back pain.

Hypothesis: We hypothesize that our active mindfulness-based meditation intervention will be feasible and acceptable to community-dwelling older adults with chronic low back pain and improve pain and symptoms to a greater extent than older adults randomized to a sham mindfulness-based meditation group.

Aim 2: to test the effect of the mindfulness-based meditation intervention on the host Gut-Brain Axis (GBA).

Hypothesis: We hypothesize that older adults randomized to the active mindfulness-based meditation intervention will have significantly improved compositional patterns and functional profiles of gut microbiota and increased pain-related cortical response measured by functional near-infrared spectroscopy (fNIRS) to a greater extent than older adults randomized to the sham mindfulness-based meditation group at 2-weeks post-intervention, and 8-weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

1. aged 50 years older
2. intact cognition (examined by the Mini-Mental State Exam, ≥ 24)
3. experiencing moderate low back pain daily or almost every day at least the previous three months (≥3 out of 10 on numeric rating scale [NRS])
4. able to speak and read English
5. not intent to change medication regimens for pain throughout the trial

Exclusion Criteria:

1. serious underlying illness (e.g., malignant neoplasms, bloodborne illness, low blood platelet count, been in chemotherapy)
2. psychosis
3. function limitation precluded the meditation practice
4. participated meditation program before
5. no access to the internet

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity and interference | Baseline and 2 weeks and 8 weeks
  Pain Inventory (BPI) will be used to assess the multidimensional aspects of pain, its location, intensity, and interference. A higher score indicated higher pain intensity with 0 indicating no pain and 10 indicating the worst pain. A higher score of pain interference means daily functions are more impacted by pain, and 0 indicates no pain interference, and 10 means the worst pain interference.

SECONDARY OUTCOMES:
Change in pain sensitivities | Baseline and 2 weeks and 8 weeks
  Quantitative sensory testing (QST) will be used to measure sensitivity to experimental pain with standardized stimuli to test both nociceptive and non-nociceptive systems.
Change in pain modulation | Baseline and 2 weeks and 8 weeks
  Conditioned pain modulation (CPM) will also be measured. The CPM effect will be calculated as the pressure pain threshold difference between the rating at the initiation and the rating at the 60 seconds of the cold stimuli.
Change in chronic pain self-efficacy | Baseline and 2 weeks and 8 weeks
  Chronic Pain Self-Efficacy Scale (CPSES) will be used to measure pain self-efficacy with scores from 0-100, higher scores indicating improved self-efficacy.
Change in anxiety | Baseline and 2 weeks and 8 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) profile will be used to measure the co-occurring anxiety. The T-score of PROMIS measurement ranges from 0 to 100 and a higher T-score indicates a more severe symptom reported by the subjects. A T-score greater than 50 means participants have more severe symptoms than the healthy population.
Change in depression | Baseline and 2 weeks and 8 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) profile will be used to measure the co-occurring depression. The T-score of PROMIS measurement ranges from 0 to 100 and a higher T-score indicates a more severe symptom reported by the subjects. A T-score greater than 50 means participants have more severe symptoms than the healthy population.
Change in fatigue | Baseline and 2 weeks and 8 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) profile will be used to measure the co-occurring fatigue. The T-score of PROMIS measurement ranges from 0 to 100 and a higher T-score indicates a more severe symptom reported by the subjects. A T-score greater than 50 means participants have more severe symptoms than the healthy population.
Change in sleep disturbance | Baseline and 2 weeks and 8 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) profile will be used to measure the co-occurring sleep disturbance. The T-score of PROMIS measurement ranges from 0 to 100 and a higher T-score indicates a more severe symptom reported by the subjects. A T-score greater than 50 means participants have more severe symptoms than the healthy population.
Change in pain-related cortical response | Baseline and 2 weeks and 8 weeks
  Cortical activity associated with pain stimuli will be assessed utilizing a continuous-wave, multichannel functional near-infrared spectroscopy (fNIRS) imaging system (LIGHTNIRS, Shimadzu, Kyoto, Japan) equipped with three semiconductor lasers emitting at 780, 805, and 830 nm. Optical data will be gathered while subjects undergo thermal pain stimulation.
Measurement and comparison of fecal microbiota alpha diversity, beta diversity, and abundance of microbial taxa in the human gut | Baseline and 2 weeks and 8 weeks
  The 16S rRNA V4 region will be amplified and sequenced by using stool samples to depict the fecal microbiota alpha diversity, beta diversity, and abundance of microbial taxa in the human gut.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be available upon reasonable request. Requests to access these datasets should be directed to jc22db@fsu.edu.